CLINICAL TRIAL: NCT03162432
Title: High Dose Interval Vitamin D Supplementation in Patients With IBD Receiving Remicade
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Web, Assistant Professor of Pediatrics, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND 135093
Record Dates: First submitted 2017-05-15; First posted 2017-05-22 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: IBD; Ulcerative Colitis; Crohn Disease
Keywords: IBD
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vitamin D3 Treatment (Experimental): Subjects receiving Remicade will be treated with oral Vitamin D3
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Oral Vitamin D3 therapy.

SUMMARY:
The goal of this study will be to assess the safety and efficacy of high-dose interval Vitamin D3 therapy in children and young adults with Inflammatory Bowel Disease being treated with serial Remicade infusions.

DETAILED DESCRIPTION:
Study subjects will receiving 50,000 units of Vitamin D3 if they receive Remicade infusions every 4-6 weeks. Study subjects will receiving 100,000 units of Vitamin D3 if they receive Remicade infusions every 6-8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Existing diagnosis of IBD
* Age 0-25 years
* Measured serum level of 25-OH Vitamin D of 15-29 ng/ml in the last 8 weeks and no changes in Vitamin D supplementation in the interim

Exclusion Criteria:

* Pregnant Women
* History of underlying kidney disease
* History of granulomatous disease
* Inability to take oral Vitamin D
* History of hypercalcemia or hypercalciuria
* Currently taking an anti-epileptic medication
* History of pre-existing liver disease (excluding primary sclerosing cholangitis, non-alcoholic fatty liver disease, or steatohepatitis)

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Ability of intervention to maintain 25-OH Vitamin D levels in the 35-80 range | Patients will continue to receive oral Vitamin D therapy for one year. We will be assessing the efficacy of oral Vitamin D therapy, in this dosing schema, to result in 25-OH Vitamin D levels during and at the conclusion of this one-year study.
  The study will involve measuring serum 25-OH Vitamin D levels after the initiation of open-label therapy. This will be done approximately one month after starting therapy, at the end of the study interval (one year), and as clinically indicated over the course of the year. Serum 25-OH Vitamin D levels are the most robust metric for assessing Vitamin D sufficiency.

SECONDARY OUTCOMES:
Assess risk of kidney stones development in patients treated with high-dose interval Vitamin D | Patients will be monitored for urinary symptoms and complete serial urine assessments as outlined in the protocol. The impact of oral Vitamin D administration on calcium excretion will be evaluated during and at the conclusion of this one-year study.
  Patients will provide a spot urine collection the day prior to their Remicade infusion. A second spot urine collection will be collected on the day of the infusion. Urinary calcium excretion will be assessed. Changes in urinary calcium excretion will be used to identify subjects at risk for the development of renal stones.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gordon RJ, Wells R, Johansen C, Liu S, Dahlberg SE, Snapper SB, Rufo PA. Efficacy and Safety of High-dose Cholecalciferol in Patients With Inflammatory Bowel Disease Receiving Infliximab. J Pediatr Gastroenterol Nutr. 2022 Apr 1;74(4):476-483. doi: 10.1097/MPG.0000000000003386. Epub 2022 Jan 18. PMID 35045559